CLINICAL TRIAL: NCT03750630
Title: A Pilot Survey to Establish Vision Health Surveillance Indicators for Children and Adolescent in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201510078RINB
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-03

CONDITIONS: Vision Status
Keywords: vision, children, adolescent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research project is to develop a vision surveillance system, in order of understanding the vision health status of children and adolescents in Taiwan.

DETAILED DESCRIPTION:
The purpose of this research project is to develop a vision surveillance system, in order of understanding the vision health status of children and adolescents in Taiwan. It can serve as a basis for the government to establish a nationwide vision surveillance system, invest research resources, and make national policies.

This research project also classified the urbanization of sampling school as high, medium and low based on the location of school.This research project explored and analyzed the health status of myopic schoolchildren and associated factors such as families, genetics, school environment, living environment and behaviors among north, south, west and east regions of Taiwan.

ELIGIBILITY:
Inclusion Criteria:

- Students with age between 3 to 18 years old

Exclusion Criteria:

1. Students have any special ocular disease.
2. non-compliance with screening protocol
3. orthokeratology user

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Students with age between 3 to 18 years old
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Refractive status | 1 day
  Cycloplegic spherical refraction measured by auto-refractometer (Diopter) in children and adolescents.

SECONDARY OUTCOMES:
Axial length | 1 day
  The axial length is the distance between the anterior surface of the cornea and the fovea and is the primary determinant of non-syndromic myopia. In this research project, investigators measure the axial length in children and adolescents by A-scan.
Intraocular pressure | 1 day
  Intraocular pressure is the pressure created by the continual renewal of fluids within the eye. In this research project, investigators measure the intraocular pressure in children and adolescents by Icare Tonometer.
Corneal thickness | 1 day
  Corneal thickness is an important factor in accurately diagnosing eye pressure. In this report project, investigators measure the corneal thickness in children and adolescents by A-scan.
Fundus examination | 1 day
  The fundus is the portion of the inner eye that can be seen during an eye examination by looking through the pupil. In this research project, investigators perform the fundus examination in children and adolescents by ophthalmoscope.
Serious and non-Serious Adverse Events | 1 day
  The adverse events in children and adolescents
Questionnaire | 1 day
  Associated factors such as families, genetics, school environment, living environment and behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan